CLINICAL TRIAL: NCT06118541
Title: To Investigate the Effects of Vestibular Rehabilitation Exercise on Dizziness, Body Balance, Post Concussion Syndrome, Anxiety and Quality of Life in Patients With Mild Traumatic Brain Injury
Brief Title: Vestibular Rehabilitation Exercise in Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202203063RINB
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Vestibular Rehabilitation
Keywords: Traumatic Brain Injury; Vestibular Rehabilitation therapy; Dizziness; Quality of Life
MeSH Terms: conditions — Brain Injuries, Traumatic; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation therapy (Experimental): The experimental group received a "vestibular rehabilitation exercise" program, The assessment tools used in this study included the Chinese version of the Dizziness Handicap Inventory (DHI), Dizziness Visual Analog Scale (DVAS), 16-item Post-Concussion Symptom Checklist (PCSC), Beck Anxiety Inventory (BAI), Traumatic Brain Injury Quality of Life (TBI-QOL) questionnaire, and a standing balance test. Measurements were taken at baseline and at weeks 2, 4, 8, and 12 post-intervention
  Interventions: Behavioral: Vestibular Rehabilitation therapy
- standard care (Experimental): Monitor the patient's consciousness and limb muscle strength, give drugs according to the time point of administration, and educate the importance of early getting out of bed
  Interventions: Behavioral: Vestibular Rehabilitation therapy

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation therapy — Vestibular rehabilitation exercises of 30 to 60 minutes twice a week for eight weeks
  Vestibular rehabilitation exercise program:
  1. Eye-Head Coordination exercise
  2. Sitting balance exercises
  3. Standing Static balance exercises
  4. Standing Dynamic balance exercises
  5. Ambulation exercises

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of long-term disability and mortality. The costs associated with hospitalization, rehabilitation, and productivity losses after injury impose a significant socioeconomic and healthcare burden. TBI patients often struggle with symptoms such as dizziness and post-concussion syndrome, preventing them from returning to their previous level of functioning. This leads to negative consequences, including unemployment, psychosocial adjustment difficulties, and decreased quality of life, particularly affecting young working-age individuals.

The purpose of this study was to investigate whether vestibular rehabilitation exercises for mild traumatic brain injury (mTBI) patients could improve symptoms of dizziness, post-concussion syndrome, physical balance, anxiety, and quality of life. The study aimed to provide individualized care plans for mTBI patients, reducing symptom burden, lowering healthcare costs, and enhancing their quality of life.

DETAILED DESCRIPTION:
This research employed a single-blind randomized clinical trial design. Participants were recruited from a teaching hospital in the central region of Taiwan, including patients from the neurosurgery ward, emergency department, and outpatient clinics. The experimental group received a "vestibular rehabilitation exercise" program, while the control group received "standard care." The assessment tools used in this study included the Chinese version of the Dizziness Handicap Inventory (DHI), Dizziness Visual Analog Scale (DVAS), 16-item Post-Concussion Symptom Checklist (PCSC), Beck Anxiety Inventory (BAI), Traumatic Brain Injury Quality of Life (TBI-QOL) questionnaire, and a standing balance test. Measurements were taken at baseline and at weeks 2, 4, 8, and 12 post-intervention. Data analysis included descriptive statistics and inferential statistics, such as independent sample t-tests, chi-square tests, Pearson's correlation coefficient, Fisher's exact test, and generalized estimating equations.

A total of 70 mTBI patients were enrolled in this study, with an average age of 54.40 (±20.43) years. The majority were male (62.80%), and the average time from injury to vestibular rehabilitation exercise initiation was 2.4 days. The two groups did not differ significantly in terms of age, gender, employment status, economic status, marital status, TBI history, cause of injury, or chronic illnesses (p > 0.05), except for education level (p = 0.005). There were no significant differences in the DHI, DVAS, immediate standing balance test, and PCSC scores between the two groups (p > 0.05) at baseline. However, significant differences were observed in anxiety levels (p = 0.032) and quality of life (p = 0.030). Results revealed the following: Dizziness: Both groups showed significant improvements in DHI and DVAS scores over time (p < 0.001), indicating that dizziness symptoms gradually improved. The experimental group demonstrated significantly better improvements in DHI and DVAS scores at weeks 2, 4, and 8 (p < 0.05), suggesting that vestibular rehabilitation exercises were more effective in reducing dizziness symptoms compared to standard care. Post-Concussion Syndrome: Both groups exhibited significant reductions in PCSC scores over time (p < 0.001), indicating gradual improvement in post-concussion symptoms. However, the experimental group showed a significant group and time interaction effect at week 4 (p = 0.033), indicating better improvement in post-concussion syndrome symptoms compared to the control group. Physical Balance: Both groups demonstrated significant improvements in standing balance (standing time) over time (p < 0.001). The experimental group exhibited significant group and time interaction effects at weeks 4, 8, and 12 (p < 0.01), indicating better improvement in physical balance (increased standing time) compared to the control group. Quality of Life: Both groups showed significant improvements in quality of life scores over time (p < 0.001). The experimental group exhibited significant group and time interaction effects at weeks 4, 8, and 12 (p < 0.001), indicating better improvement in quality of life compared to the control group. Anxiety: Both groups demonstrated significant reductions in anxiety scores over time (p < 0.001). The experimental group exhibited significant group and time interaction effects at weeks 2, 4, 8, and 12 (p < 0.01), indicating greater reduction in anxiety symptoms compared to the control group.

In conclusion, vestibular rehabilitation exercises can reduce dizziness, alleviate post-concussion syndrome, improve physical balance, reduce anxiety, and enhance the quality of life in mTBI patients. It is recommended to extend the implementation of these exercises to other hospitals to benefit patients with similar symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Within 2 weeks of diagnosis of mild head trauma (mild TBI, mTBI).
2. Adults over 20 years old
3. Coma Index (GCS) ≧ 13 points in the emergency department
4. Those who have three or more symptoms using the concussion syndrome checklist
5. No visual or hearing impairment
6. No fractures, no movement, mental illness and central related diseases
7. No cognitive impairment 8. Agree to participate in this study

Exclusion Criteria:

1. Patients with mental disorders and cognitive dysfunction
2. Those who relied on others for assistance in daily living activities prior to injury
3. Patients who have been diagnosed with inner ear disease causing balance problems
4. Patients who have been diagnosed with anxiety disorders before the injury

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | The measurement time points were the time of receipt and the 2nd, 4th, 8th, and 12th weeks after intervention
  The self-perception impairment of vestibular system disorders is assessed into three categories, representing "dizziness and unstable functioning", "emotional" and "physical", with a "yes", "no" or "sometimes" response to each item scoring 4 points; 2 points for responding to "sometimes"; and response "no" 0 points. The total score ranges from 0 (accessibility) to 100 (maximum score), with a total score between 0 and 50 indicating occasional dizziness, 51 to 60 indicating frequent dizziness and 61 to 100 indicating persistent dizziness
Dizziness Visual Analog Scale (DVAS) | The measurement time points were the time of receipt and the 2nd, 4th, 8th, and 12th weeks after intervention
  Draw a 100mm straight line, 0 cm on the far left, 10 cm on the far right, 0 means no dizziness, 10 means the dizziness is very severe, if the score is between 1-4 cm means mild dizziness, 4-8 cm means moderate dizziness, and between 8-10 cm is severe dizziness, take a pen and ask the patient to draw an X vertically on this straight line, representing the degree of his dizziness, and then use a ruler to measure the value and record it
The 5 times sit to stand test(FTSTS) | The measurement time points were the time of receipt and the 4th, 8th, and 12th weeks after intervention
  The patient is asked to be able to sit independently in a chair without armrests, with his hands crossed over his chest, to stand and sit down 5 times as soon as possible, and to record the time of completion
16-item Post-Concussion Symptom Checklist (PCSC) | The measurement time points were the time of receipt and the 2nd, 4th, 8th, and 12th weeks after intervention
  including Headache, dizziness, nausea, vomiting, tinnitus, blurred vision, tiredness, poor physical strength, sleep disturbances, memory impairment, unresponsiveness, depression, irritability, difficulty concentrating, and other symptoms. The CPCS is divided into two parts: pre-injury and post-injury, before the injury is asked whether there are 16 symptoms, if there are any, the severity of the symptoms is assessed, and the Likert Scale 5-point (0-4) score is used to compare the problem symptoms with the situation before the head injury, 0 points means "not at all", 1 point means "mild", 2 points means "moderate", 3 points means "severe", 4 points indicate "very severe", the total score is 0-64 points, the higher the score, the more severe the symptoms. After the injury, the Likert Scale was used to score 5 points (1-5), 1 point means "significantly mild", 2 points means "slightly mild", 3 points indicate "unchanged", 4 points indicate
Beck Anxiety Inventory(BAI) | The measurement time points were the time of receipt and the 2nd, 4th, 8th, and 12th weeks after intervention
  The patient self-assessed the level of anxiety in the past week, with the highest score of 3 and the lowest score of 0 for each question, and the score of "not at all" was 0. 1 point for "slight"; 2 points for "frequently occurring"; A score of 3 is given for "severe", with a total score ranging from 0-63, with 0-7 being "normal", 8-15 being "mild anxiety", 16-25 being "moderate anxiety" and 26-63 being "severe anxiety"
Quality of Life after Brain Injury(QOLIBRI) | The measurement time points were the time of receipt and the 4th, 8th, and 12th weeks after intervention
  Applicable to traumatic brain injury and at all points in time after injury, it consists of 37 items in 2 parts, 6 aspects of satisfaction, including cognition, self (including, e.g., energy, motivation, self-esteem, self-perception), daily life and autonomy, social relationships, emotions, and physical problems. The first part assesses the patient's four aspects: cognition (7 items), self (7 items), daily life and autonomy (7 items), and social relationships (6 items), while the second part assesses two aspects: emotions (5 items) and physical problems (5 items). The Likert Scale is scored on a 5-point scale (1-5), ranging from 1 (no distress at all) to 5 (very distressed), in which emotional and physical conditions are inversely scored, with higher total scores indicating higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chun Liao, Principal Investigator — National Taiwan Hospital Yunlin Branch; Pei-Yin Sun, Principal Investigator — National Taiwan Hospital Yunlin Branch
Locations (1):
- National Taiwan Universiyt Hospital Yunlin Branch, Yuanlin, Taiwan